CLINICAL TRIAL: NCT04895020
Title: Evaluating the Immunogenicity and Safety of 9-valent Human Papillomavirus(Type6, 11, 16, 18, 31, 33, 45, 52 and 58) Recombinant Vaccine in Chinese Females Aged 9 to 45 Years: A Phase 3, Open-label, Non-randomised Clinical Trial
Brief Title: Immunobridging Study of 9-valent Human Papillomavirus Recombinant Vaccine in Chinese Females Aged 9 to 19 Years
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Bovax Biotechnology Co., Ltd. (Industry)
Collaborators: Chongqing Bovax Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 9-HPV-3003
Record Dates: First submitted 2021-05-17; First posted 2021-05-20 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: HPV Infections; Cervical Cancer; Vulvar Cancer; Vaginal Cancer; CIN1; CIN2; CIN 3; VaIN1; VaIN2; VaIN3; Genital Wart; VIN 1; VIN 2; VIN 3; AIS
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms; Vulvar Neoplasms; Vaginal Neoplasms; Condylomata Acuminata

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 9-valent HPV vaccine (Experimental): 9-valent HPV recombinant vaccine (Hansenula Polymorpha) All subjects aged 9 to 45 years received 3 doses of 9v HPV vaccine at 0,2,6 month scehdule
  Interventions: Biological: 9-valent HPV vaccine

INTERVENTIONS:
Biological: 9-valent HPV vaccine — 9-valent HPV recombinant vaccine (Hansenula Polymorpha) All subjects aged 9 to 45 years received 3 doses of 9v HPV vaccine at 0,2,6 month scehdule

SUMMARY:
This phase 3 study will evaluate the immunogenicity and safety of 9-valent HPV recombinant vaccine in Chinese females aged 9 to 45 years

DETAILED DESCRIPTION:
This study (protocol 9-HPV-3003) is an immunogenicity and safety study in the subjects (9-19 years of age) who received the 9-valent HPV recombinant vaccine compared with the subjects (20-45 years of age). In this study, we will assess whether the immunogenicity of the 9-valent HPV vaccine given 3-dose schedule in the subjects (9-19 years of age) in noninferior to that in the subjects (20-45 years of age) receiving 3 doses, while assessing the safety of this vaccine.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for the first stage:

1. Healthy Chinese females aged 9 to 45 years; Provide legal identification;
2. The subject voluntarily agrees to enroll in this study. If the subject is a minor, both the subject and subject's legal guardian should voluntarily agree to enroll in this study and sign an informed consent form;
3. Be able to understand the study procedures and promise to participate in regular follow-ups under the requirements;
4. Had a negative urine pregnancy test on the day of enrollment, among the subjects of childbearing age; Not in the duration of breast-feeding and no birth plan within 7 months; According to the investigator's judgment that there is no possibility of pregnancy at that time: subjects have taken effective contraception, or asexual life after the last menstrual period, or use IUD, or had undergone ligation; subjects agree to continue take effective contraception such as taking OCS and condom use;
5. No fever symptoms on the day of enrollment (aged> 14 years old, axillary temperature<37.3°C; aged ≤ 14 years old, axillary temperature<37.5°C );

   Inclusion Criteria for the second stage:
6. Received all 3 doses of trial vaccination;
7. Subjects aged 9 to 19 years at the first stage.

Exclusion Criteria:

1. Received marketed HPV vaccine or plan to receive marketed HPV vaccine during this study period or have enrolled in HPV vaccine clinical trials;
2. History of positive test to HPV, history of cervical cancer (e.g. abnormal screening test results, abnormal cervical biopsy results, including CIN, AIS, and cervical cancer) or history of hysterectomy (vaginal or abdominal radical hysterectomy), or history of pelvic radiotherapy; History of genital diseases related to HPV infection (e.g. uterine peristalsis, VIN, VAIN, AIN, and related cancers); History of STDs, including syphilis, gonorrhea, genital herpes, Mycoplasma genitalium, Lymphgranuloma Venereum, granuloma inguinale, etc.;
3. Known allergy to any vaccine components or history of severe allergic diseases requiring treatment, including shock, laryngeal edema, urticarial, Henoch-Schonlein purpura, Arthus reaction, etc.;
4. Had primary or acquired immunodeficiency such as HIV, SLE, JRA, etc. or received immunosuppressive treatment within one month before study such as long-term glucocorticoid use(≥2mg per kg per day, lasted more than two wks), or plan to receive such treatment from day 0 to month 7 after the last dose;
5. Had chronic diseases or congenital malformations, which might interfere with the process and completion of this study, such as Down Syndrome, heart diseases, liver diseases, chronic diabetes complications, and malignant tumor;
6. Enrolling or plan to enroll in other clinical trials (drug or vaccine);
7. Had infectious diseases such as TB, viral hepatitis, and/or HIV infection;
8. Had convulsions, epilepsy, encephalopathy, and mental illness or family history;
9. With prohibitive contraindications such as Thrombocytopenia or coagulopathy;
10. Asplenic, functionally asplenic, or splenectomy caused by any condition;
11. Within 3 days prior to vaccination, have an acute disease or are in the acute attack of a chronic disease or have used antipyretic, analgesic and anti-allergic drugs (such as: acetaminophen, ibuprofen, aspirin, loratadine, ceti Rizine, etc.);
12. Receipt of inactivated or recombinant vaccines within 14 days, live vaccines within 28 days;
13. Receipt of immune globulin or blood-related products within 3 months; or plan to receive such products during this study period;
14. Had fever symptoms within 24 hours on the first day (aged> 14 years old, axillary temperature ≥ 37.3°C; aged ≤ 14 years old, axillary temperature ≥37.5°C );
15. Untreated/uncontrolled hypertension before vaccination (aged 9 to 17 years: systolic BP>120mmHg and/or diastolic BP>80mmHg; aged more than 18 years: Systolic BP≥140mmHg and/or diastolic BP ≥90mmHg);
16. Plan to permanently relocate from the area before the end of the study or leave the local area for a long time during the study visit (affecting the scheduled visit time);
17. According to the investigator's judgment, the subject has any condition may interfere with process of evaluation or participating in this study cannot guarantee the object's maximum benefit.

Ages: 9 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1200 (Estimated)
Dates: Start 2021-05-28 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
The primary immunogenicity objective | 30 days after the last dose(3 doses schedule)
  The primary outcome measure for assessing vaccine immunogenicity, among subjects aged between 9 and 45, is the results of seroconversion rate of neutralizing antibodies after immunization in pre-immune negative subjects from 30 days after the last dose (3 doses schedule, Month 7) to HPV 6, 11, 16, 18, 31, 33, 45, 52 , and 58.

SECONDARY OUTCOMES:
Number of patients with postive antibodies after the whole schedule vaccination from the former negative subjects | 30 days after the last dose(3 doses schedule)
  The secondary outcome measure for assessing vaccine immunogenicity, among subjects aged between 9 and 45, is the geometric mean titer (GMT) from 30 days after the last dose (3 doses schedule, Month 7) to HPV 6, 11, 16, 18, 31, 33, 45, 52 , and 58.
Rate of seroconversion among the patient aged 9-26 after the whole schedule vaccination | 30 days after the last dose(3 doses schedule)
  To assess vaccine immunogenicity among the subjects aged between 9 and 26, is the seroconversion rate of neutralizing antibodies and the GMT from 30 days after the last dose (3 doses schedule, Month 7) to HPV 6, 11, 16, 18, 31, 33, 45, 52 , and 58.
GMT and seropositive rate of HPV in the 9-19 age group after 60-month follow-up | Day 1 to 60 months post vaccination 3
  After receiving all 3 doses vaccinations, the subjects aged 9 to 19 years will be followed for 60 month (Month 12/24/36/48/60) after first vaccination to assess the GMT and seropositive rate (4-fold-increase) to HPV 6, 11, 16, 18, 31, 33, 45, 52, and 58.

OTHER OUTCOMES:
Number of AE within 30 minutes after each dose | 30 mins after each dose
  Adverse events reported within 30 minutes after each dose
Number of SAE within 7days after each dose | day 0 to day 7 after each dose
  Solicited adverse events reported between day 0 to day 7 after each dose
Number of unsolicited adverse events within 30days after each dose | day 0 to day 30 after each dose
  Unsolicited adverse events reported between day 0 to day 30 after each dose
Number of all SAE during the study period | Stage 1: from month 6 to month 12 after the last dose; Stage 2: 6 month after receiving the whole vaccine schedule to 60 month after the 1st dose
  Serious adverse events reported during the study period
Number and rate of pregnancy events | Stage 1: from month 6 to month 12 after the last dose; Stage 2: 9-to-19-year-old subjects received 3 doses vaccinations, 6 month after receiving the whole vaccine schedule to 60 month after the 1st dose
  Pregnant event and pregnant outcome reported during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Person(s) responsible for the overall scientific leadership of Lv, Study Director — Zhejiang Provincial Center for Disease Control and Prevention
Locations (1):
- Huakun Lv, Hangzhou, China